CLINICAL TRIAL: NCT03742154
Title: A Pilot Translational Study of Varenicline Sampling to Promote Treatment Engagement and Smoking Cessation
Brief Title: Hollings Cancer Center Varenicline Sampling Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Matthew Carpenter, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00078289
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Smoking; Smoking Cessation; Smoking, Tobacco; Smoking, Cigarette
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Smoking; Cigarette Smoking | interventions — Varenicline

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of the two study groups, like drawing numbers from a hat. One group will receive a mailed sample of varenicline, and the other will not. Participants have 50/50 chance of being in either group. Both groups will contain equal numbers of smokers motivated to quit and smokers not currently motivated to quit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Varenicline Group (Experimental): 50 participants will be enrolled in this group. They will receive a sample of varenicline to use for up to 4-weeks. They are receiving 40 - 0.5mg pills of varenicline, with instructions for titration.
  Interventions: Drug: Varenicline 0.5 MG
- Control Group (No Intervention): 49 participants will be enrolled in this group.

INTERVENTIONS:
Drug: Varenicline 0.5 MG — varenicline comes in bottles of 56 - 0.5 mg pills
  Other Names: Chantix; Varenicline Pill
  Arms: Varenicline Group

SUMMARY:
The purpose of this study is to learn what happens when people are given a free, 4-week, sample of varenicline, a smoking cessation medication. Investigators will look at quit attempts, changes in smoking, and attitude towards varenicline, in both smokers who want to quit and those who do not.

Smoking use causes a number of deaths and diseases, including heart disease and cancer. All smokers are advised to quit. Varenicline (sometimes called Chantix), is a prescription medication approved by the US FDA. Many studies show that use of varenicline can help smokers quit smoking.

Varenicline is a prescription medication, which usually means that people have to see a doctor to get it. This study examines a different way to deliver varenicline, delivered directly to participants for a few weeks, and without need to see a doctor. This method is called "varenicline sampling."

The study is sponsored by the Hollings Cancer Center at the Medical University of South Carolina. The study is being done at the Medical University of South Carolina, but study recruitment is based state-wide, throughout South Carolina.

ELIGIBILITY:
Inclusion Criteria:

* age 18+
* daily smoker (25+ days/previous month)
* smoking 5+ cigarettes/day;
* smoking > 1yr;
* some interest in eventual quitting (>2 on 10-point scale);
* has a primary care doctor and has seen that doctor at least once in past year; and
* own a smartphone or have regular (daily) access/use of email.

Exclusion Criteria:

* reports of history of seizures or seizure disorders;
* suicidal ideation in past month;
* any lifetime suicide attempt;
* currently pregnant, breastfeeding, or planning to become pregnant; or
* reports of hallucinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carpenter MJ, Gray KM, Wahlquist AE, Cropsey K, Saladin ME, Froeliger B, Smith TT, Toll BA, Dahne J. A Pilot Randomized Clinical Trial of Remote Varenicline Sampling to Promote Treatment Engagement and Smoking Cessation. Nicotine Tob Res. 2021 May 24;23(6):983-991. doi: 10.1093/ntr/ntaa241. PMID 33249458

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varenicline Group | Control Group
Started | 50 | 49
Completed | 50 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Group: 50 participants will be enrolled in this group.
- Total: Total of all reporting groups
Arm/Group | Varenicline Group | Control Group | Total
Number analyzed (Participants) | 50 | 49 | 99
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.0 (12.8) | 40.4 (11.5) | 41.7 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 35 | 57
  Male | 28 | 14 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 40 | 35 | 75
  Black | 8 | 10 | 18
  Multiracial | 2 | 3 | 5
  American Indian or Alaska Native | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 50 | 49 | 99
Baseline Cigarettes Per Day (7 day avg) [Mean (Standard Deviation); unit: cigarettes per day] | 18.4 (7.2) | 15.1 (7.3) | 16.8 (7.3)
Cigarette Dependence (Heaviness of Smoking Index) [Mean (Standard Deviation); unit: units on a scale] — Scale of 0-6 where 0 is lowest addiction and 6 is highest addiction.
  units on a scale | 3.4 (1.3) | 2.8 (1.5) | 3.1 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Quit Attempts
Description: Percent of participants with any self-defined and any self-defined 24-hr quit attempt
Time Frame: From study enrollment through end of three-month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline Group | Control Group
Number analyzed (Participants) | 50 | 49
Participants
  Any self defined quit attempt | 30 | 24
  Any 24 hour quit attempt | 26 | 17

2. Secondary Outcome: Conversion of Varenicline Use
Description: Percent of participants in the sampling group using varenicline at 3-month follow up assessment.
Time Frame: At the end of the three-month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline Group
Number analyzed (Participants) | 50
Participants
  Any use of varenicline | 12
  Daily use of varenicline | 5

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | Varenicline Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 26/50 | 10/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline Group (N=50) | Control Group (N=49)
Sleep Disturbance (General disorders) | 16 | 3
Insomnia (General disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 11 | 1
Agitation (General disorders) | 7 | 1
Depressed Mood (General disorders) | 5 | 2
Headache (General disorders) | 4 | 5
Constipation (Gastrointestinal disorders) | 3 | 0
Gas (Gastrointestinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT03742154/Prot_SAP_000.pdf